CLINICAL TRIAL: NCT03337126
Title: A Phase 1, Randomized, Open-Label, Single Dose, Two Sequence, Crossover, Relative Bioavailability and Taste Test Study of ATI-1501 in Healthy Adult Volunteers
Brief Title: Bioavailability of ATI-1501 With Taste Test Sub Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Appili Therapeutics Inc. (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ATI-1501-02
Record Dates: First submitted 2017-11-06; First posted 2017-11-08 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Bioequivalence
MeSH Terms: interventions — Metronidazole

STUDY DESIGN:
Intervention Model Description: Randomized, Open-Label, Single Dose, Two Sequence, Crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fasting Condition (Active Comparator): Single dose of ATI-1501(oral suspension) administered under fasting conditions; BioAvailability and PK parameters will be measured and analyzed. These parameters will be compared to the BA and PK parameters measured after administration of a single Metronidazole Tablet
  Interventions: Drug: Metronidazole Tablet
- Fed Condition (Active Comparator): Single dose of ATI-1501(oral suspension) administered under fed condition; BioAvailability and PK parameters will be measured and analyzed. These parameters will be compared to the BA and PK parameters measured after administration of a single Metronidazole Tablet
  Interventions: Drug: Metronidazole Tablet

INTERVENTIONS:
Drug: Metronidazole Tablet — Comparator Drug
  Other Names: Flagyl

SUMMARY:
Appili Therapeutics Inc. is developing an oral suspension formulation of metronidazole (ATI-1501), a taste-masked reformulation of metronidazole. The purpose of this study is to compare the relative bioavailability of ATI-1501 with the Reference Listed Drug (RLD) in healthy, adult volunteers to determine that it is Bioequivalent.

DETAILED DESCRIPTION:
This is a Phase 1, single-center, randomized, open-label, single dose, 2 sequence, 2 treatment, crossover, relative bioavailability study of ATI-1501 under fasting and fed conditions in healthy adult subjects. The purpose of this study is to determine the relative bioavailability of ATI-1501 oral suspension to the comparator drug, Flagyl®. The study also aims to evaluate the safety and characterize the PK profile of ATI-1501 oral suspension in healthy adults. The PK of ATI-1501 oral suspension in a population of subjects with no concomitant illnesses will be recorded and analyzed. Blood samples will be collected through individual venipuncture or an indwelling catheter at pre-described time intervals throughout the study to determine the bioavailability of ATI-1501 oral suspension and characterize its overall PK profile. In addition, blood samples will also be collected using a microsampling device to validate the use of blood microsampling for future studies. Subjects will be randomized to 1 of 2 treatment sequences and each group of subjects will undergo 4 periods of treatment. Each subject will receive each treatment regimen in this crossover study design, allowing for a 7-day washout period. The study drugs will be administered under fasting and fed conditions to evaluate the effects of food on the absorption of metronidazole, administered in the ATI-1501 oral suspension. The palatability of ATI-1501 will be assessed using the 9-point scale to assess the taste, texture, and smell of the 2 study drugs. A 3-point scale will be used to evaluate the degree of bitterness of the 2 study drugs

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects 18 to 65 years of age, inclusive.
2. Body mass index (BMI) within the range of 18.0 to 30.0 kg/m2, inclusive, and a minimum weight of 50.0 kg.
3. Continuous non-smoker for at least 3 months prior to screening and tests negative on urine cotinine confirmatory test.
4. Female subjects of childbearing potential with male sexual partners must be using and willing to continue using medically acceptable contraception for at least 1 month prior to screening (at least 3 months for oral and transdermal contraceptives) and for at least 1 month after the last study drug administration.
5. Female subjects of non-childbearing potential
6. Male subjects with female sexual partners of childbearing potential must be using and willing to continue using medically acceptable contraception from screening and for at least 1 month after the last study drug administration.
7. Able to speak, read, and understand English sufficiently to allow completion of all study assessments.
8. Must provide written informed consent prior to the initiation of any protocol-specific procedures.

Exclusion Criteria:

1. History or presence of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or influence the results of the study, such as evidence of gastrointestinal (GI), hepatic or renal disease that may affect absorption, distribution, metabolism, or excretion of the orally administered study drug.
2. Recent history (within 4 weeks prior to screening) or current active infection associated with fever and/ or requiring antibiotic therapy.
3. Presence of latent or chronic infection (eg, recurrent sinusitis, urinary tract infection, genital or ocular herpes).
4. Any medical/surgical procedure or trauma within 4 weeks of the first study drug administration.
5. Any malignancy within the previous 5 years, with the exception of superficial skin cancer treated with local therapy.
6. Self-reported history of substance or alcohol dependence (excluding nicotine and caffeine) within the past 2 years, and/or has ever participated or plans to participate in a substance or alcohol rehabilitation program to treat their substance or alcohol dependence.
7. Self-reported family history of substance abuse in an immediate family member (eg, parent, sibling or child).
8. Positive urine drug screen.
9. Positive breath alcohol test.
10. History or presence of clinically significant abnormality as assessed by physical examination, medical history, ECGs, vital signs, or laboratory values, which, in the opinion of the investigator, would jeopardize the safety of the subject or the validity of the study results.
11. Evidence of clinically significant hepatic or renal impairment including alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >1.5 x upper limit of normal (ULN), or bilirubin >1 x ULN.
12. Inability to fast for a minimum of 14 hours.
13. Positive for hepatitis A, hepatitis B, hepatitis C, human immunodeficiency virus (HIV) or tuberculosis.
14. Donation or loss of more than 500 mL whole blood within 30 days preceding entry into the Treatment phase.
15. Plasma donation within 7 days prior to dosing of study drug.
16. Difficulty with venous access or unsuitable or unwilling to undergo catheter insertion.
17. Female subjects who are currently pregnant (have a positive pregnancy test) or lactating or who are planning to become pregnant within 30 days of last study drug administration.
18. History of severe allergic reaction (including anaphylaxis) to any substance, or previous status asthmaticus.
19. History of allergy or hypersensitivity to Flagyl®, ATI-1501, or other nitroimidazole derivatives.
20. Subject is mentally or legally incapacitated or has significant emotional problems at the time of screening visit or expected to during the conduct of the study.
21. Use of a prohibited medication, as specified in Section 4.4.1.
22. Treatment with an investigational drug within 30 days (if the elimination half-life is unknown) prior to first drug administration or is concurrently enrolled in any research judged not to be scientifically or medically compatible with this study.
23. An employee of the sponsor or research site personnel directly affiliated with this study or their immediate family member defined as a spouse, parent, child, or sibling, whether biological or legally adopted.
24. A subject who, in the opinion of the investigator or designee, is considered unsuitable or unlikely to comply with the study protocol for any reason.
25. A subject who has pending legal charges or is on probation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2017-12-13 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Relative bioavailability | 48 hours
  Relative bioavailability of ATI-1501 compared to Flagyl® tablets under fasting and fed conditions

SECONDARY OUTCOMES:
Palatability | 4 hours
  Palatability of ATI-1501

CONTACTS AND LOCATIONS:
Overall Officials: Michael McDonnell, MD, Principal Investigator — Syneos Health
Locations (1):
- INC Research Inc., Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided